CLINICAL TRIAL: NCT04420208
Title: Ameliorating the Obstacle of Pap Smear: a Randomized Controlled Trial
Brief Title: Ameliorating the Obstacle of Pap Smear
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: 202004014RINB
Record Dates: First submitted 2020-06-04; First posted 2020-06-09 (Actual); Last update posted 2021-11-01 (Actual); Status verified 2021-10

CONDITIONS: Pain
Keywords: Cervical cancer screening; Pap smear; Procedural pain; Peak-end rule
MeSH Terms: conditions — Pain; Pain, Procedural

STUDY DESIGN:
Intervention Model Description: Subjects are divided into two groups, one with traditional Pap smear and one with Pap smear adding a non-painful procedure at the end. The investigators will compare the real-time pain score and recalled pain to check whether the theory works.
Who Masked: Participant
Masking Description: During the Pap test, there is a privacy curtain separating participants from the operators. Participants receiving the modified Pap test do not realize what is going on during the 15-second step because they are behind the privacy curtain. The operators performing the procedure are not informed whether to intervene or not by the assistants until a specimen is prepared for cervical cytology. The delayed disclosure of the group allocation until this step ensures the operators standardizing the insertion and opening phases of the Pap test.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Modified Pap test (Experimental): Adding a non-painful event after the most uncomfortable phase of Pap smear.
  Interventions: Procedure: Modified Pap test
- Traditional Pap test (No Intervention): Traditional Pap-smear procedure as control.

INTERVENTIONS:
Procedure: Modified Pap test — Adding a non-painful step after the most uncomfortable phase of Pap smear
  Arms: Modified Pap test

SUMMARY:
To reduce the procedural pain of Pap smear, this study expects to apply the peak-end rule to Pap smear by prolonging the insertion of speculum after samples are obtained from the cervix. This study aims to conduct a randomized controlled study at a tertiary center, National Taiwan University Hospital (NTUH). The investigators expect to compare the recalled pain intensity of the intervention and control groups.

DETAILED DESCRIPTION:
Purpose: In order to reduce the procedural pain, this study expects to apply the peak-end rule to Pap smear by prolonging the insertion of speculum after samples are obtained from the cervix. Methods: This study aims to conduct a randomized controlled study at NTUH. Approximately 200 subjects are expected to be recruited. The investigators will utilize the peak-end rule by adding a non-painful step right after the most uncomfortable phase in the intervention group. All study subjects are requested to score on a numeric pain scale during the Pap test. All operators experienced in techniques for performing a Pap test should attend workshops for a standard operating procedure. A well-trained research assistant is also responsible for ensuring standardization of procedures to eliminate interoperator variability. The primary outcome was the recalled pain intensity at five minutes after the Pap smear test.

ELIGIBILITY:
Inclusion Criteria:

* Biological female
* Aged 30-70
* Provision of written informed consent

Exclusion Criteria:

* Pregnancy
* Active vaginal or uterus infection
* Incapable of understanding the numeric pain scales
* Prior cervical cancer diagnosis
* Prior hysterectomy, pelvic or vaginal surgery
* Ongoing menstruation
* Use of painkillers within 24 hours

Ages: 30 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 268 (Actual)
Dates: Start 2020-05-28 (Actual); Primary Completion 2020-10-31 (Actual); Study Completion 2021-10-11 (Actual)

PRIMARY OUTCOMES:
Recalled pain just after the Pap smear test using a 1-5 numeric scale | Five minutes after the Pap test
  This recalled pain intensity is evaluated with a 1-5 numeric scale (1:no pain; 5: maximal pain).
Recalled pain just after the Pap smear test using a a 0-10 visual analog scale | Five minutes after the Pap test
  This recalled pain intensity is evaluated with a 0-10 visual analog scale (0: no pain; 10: maximal pain), where pain was categorized as mild, moderate, and severe.

SECONDARY OUTCOMES:
Real-time pain during the Pap test using a 1-5 numeric scale | Every five seconds throughout the Pap test
  The participants are asked to evaluate and record their pain every five seconds throughout the test. The real-time pain is recorded with a 1 to 5 numeric scale (1:no pain; 5: maximal) at the beginning, the first quarter, the second quarter, the third quarter, and the end of the regular course in all participants; as well as right after the additional 15-second step in the group receiving modified Pap tests. The average pain, the maximal pain, as well as real-time pain at the beginning, the first quarter, the second quarter, the third quarter, and the end of the regular course are compared between the two groups. For each group, we also compare the average pain of the first half and the second half of the total course. For participants receiving the modified Pap test, we further compare the average pain, the maximal pain, and the last recorded real-time pain of the 15-second step with that of the regular course.
Long-term recalled pain after the Pap test using a 1-5 numeric scale | One year after the Pap test
  Evaluated with a 1-5 numeric scale (1: no pain; 5: maximal pain).
Long-term recalled pain after the Pap test using a 0-10 visual analog scale | One year after the Pap test
  Evaluated with a 0-10 visual analog scale (0: no pain; 10: maximal pain).
Willingness to receive further Pap tests | One year after the Pap test
  0-10 grades (0: unwillingness; 10: highest grade of willingness)

CONTACTS AND LOCATIONS:
Overall Officials: Chien-Hsieh Chiang, MD, MPH, Study Chair — Attending physician
Locations (1):
- National Taiwan University Hosputal, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Yen HK, Cheng SY, Chiu KN, Huang CC, Yu JY, Chiang CH; NTUH Pap Study Group. Adding a nonpainful end to reduce pain recollection of Pap smear screening: a randomized controlled trial. Pain. 2023 Aug 1;164(8):1709-1717. doi: 10.1097/j.pain.0000000000002897. Epub 2023 Apr 12. PMID 37043729